CLINICAL TRIAL: NCT05606796
Title: Comparison of Preserved and Preservative-free Latanoprost 0.005% in Primary Open Angle Glaucoma and Ocular Hypertensive Patients, at Guinness Eye Centre, Lagos.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uzoma Chinyei Joan (Other)
Responsible Party: Sponsor-Investigator, Uzoma Chinyei Joan, Principal investigator, University of Lagos, Nigeria
Organization: University of Lagos, Nigeria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chinyei
Record Dates: First submitted 2022-10-24; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Randomized clinical control trial.
Who Masked: Participant, Investigator
Masking Description: Both preserved and preservative-free drugs would be masked from the patient and the principal researcher. The pharmacist would remove actual labels, and mask them with new labels, coded ''X'' and ''Y'' latanoprost 0.005%, representing either preserved or preservative free medications, known to only the pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preserved latanoprost (Experimental): Benzalkonium chloride (BAK) preserved latanoprost 0.005%.
  1 drop will be instilled into the conjunctival sac of both eyes of patient, at about 9pm daily, to reduce intraocular pressure.
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution
- Preservative-free latanoprost (Experimental): Preservative-free (Benzalkonium chloride-free) latanoprost 0.005%.
  1 drop will be instilled into the conjunctival sac of both eyes of patient, at about 9pm daily, to reduce intraocular pressure.
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: Latanoprost 0.005% Ophthalmic Solution — 1 drop of 0.005% Latanoprost (preserved or preservative-free) would be instilled into the conjunctival sac daily for 12 weeks.

SUMMARY:
It is a randomised, double-blinded clinical trial in which consenting participants who meet the inclusion criteria would be randomised into 2 groups. Subjects will be given either preserved or preservative free latanoprost for a period of 12 weeks. The efficacy and tolerability of both drugs would be assessed every 4 weeks, amongst these patients.

DETAILED DESCRIPTION:
Ethical approval has been obtained from the Health Research Ethics Committee of Lagos University Teaching Hospital.

Patients will be recruited from the weekly glaucoma clinic, Monday, Thursday, and Friday general clinics. Each participant would be seen for a period of 12 weeks; at baseline visit, and weeks 4, 8 and 12, in which topical, label-masked preserved or preservative free latanoprost would be dispensed, with patient instructed to instill one drop of 0.005% latanoprost by 9:00pm (± 1 hour). Efficacy of the two eye drops will be assessed by measuring the intraocular pressure 3 times a day at every visit. Safety and potential adverse effects of the drops will be evaluated in terms of ocular symptoms and tear parameters. Ocular symptom values of the patients will be evaluated.

All patients will undergo ocular examinations, including visual acuity assessment, slit lamp biomicroscopy, intraocular pressure, tear film breakup time (TBUT), fluorescein staining, schirmer test, gonioscopy, standard automated perimetry, and ophthalmoscopy. Tolerability will be evaluated with the frequency and percentage of distributions of severity level using the OSDI questionnaire in each group after administration at weeks 4 and 12, respectively. The symptoms checked during follow-up visits will include; pruritus, burning/stinging, blurred vision, tearing, sticky eye sensation, eye dryness sensation, and foreign body sensation. Quality of life would be evaluated at baseline visit and at week 12, using the standard quality of life Q-15 questionnaire.

A research team would be involved in carrying out this research, Comprising the principal researcher, a pharmacist, and 2 ophthalmic nurses. Results will be collated and analysed by the principal researcher. The entire research would be carried out over a period of 9 months, from December 2022 to August 2023.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed, consenting high tension, primary open angle glaucoma or ocular hypertensive patients.
* Forty years and above.
* Intraocular pressure of 21- 30mmHg (millimetres of mercury)
* Willingness to participate in the study.

Exclusion Criteria:

* Patients under 40 years of age.
* Diabetic patients
* Patients on other anti- glaucoma medications.
* Patients on topical immunosuppressive medication.
* Patients on anti-depressants.
* Patients who have had any form of ocular surgery or intervention such as cryotherapy.
* Patients using contact lens.
* Patients on any form of topical medication in the last 1 month.
* Patients diagnosed or suspected to have Sjogren syndrome.
* Patients being managed for Steven-Johnson's syndrome, ocular cicatricial pemphigoid.
* Pregnant patients.
* Previous glaucoma surgery and any refractive surgery <12 month prior to enrolment.
* Only eye patients.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure assessment. | 12 weeks
  Intraocular pressure measured in millimetre mercury (mmHg), will be assessed every 4 weeks at 8am,12pm and 4pm. Normal intraocular pressure ranges between 9 to 21mmHg. Any intraocular pressure values above 21mmHg would be considered abnormal. Pressures below 6mmHg will be considered as hypotony.

SECONDARY OUTCOMES:
Ocular surface disease index (OSDI) questionnaire. | 4 weekly in 12 weeks.
  The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patient's responses are rated on a scale of 0 to 4, with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated, which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Quality of life-15 questionnaire. | Baseline visit and week 12.
  Questionnaire is composed of 15 items, 4 domains which address factors of visual disability: central and near vision, peripheral vision, dark adaptation and glare, and outdoor mobility. Poorer QoL scores are associated with worse functional status and increased visual morbidity from glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: ADEOLA ONAKOYA, MBBS, FMCOph, FICO, Principal Investigator — Lagos State University
Locations (1):
- Guinness Eye Centre. Lagos University Teaching Hospital., Lagos, Lagos, Nigeria